CLINICAL TRIAL: NCT00133016
Title: The Efficacy of Early Amniotomy for Induction of Labor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 701340
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Labor, Induced
Keywords: Induction of labor
MeSH Terms: interventions — Amniotomy

INTERVENTIONS:
Procedure: Amniotomy

SUMMARY:
The purpose of this clinical trial is to investigate the efficacy of early amniotomy on reducing both the duration of labor and the frequency of dystocia in nulliparous women undergoing an induction of labor. This research project is a prospective, parallel clinical trial, in which subjects are randomized into one of two treatment groups: those who undergo early amniotomy and those who do not undergo early artificial rupture of the amniotic membranes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 37 weeks (using established National Institute of Child Health and Human Development [NICHD] dating criteria)
* Nulliparous (i.e., first term pregnancy)
* Admitted to the hospital for induction of labor
* Singleton pregnancy
* Fetal head applied to the cervix
* The ability to understand the requirements of the study, as determined by the study nurse

Exclusion Criteria:

* Premature rupture of amniotic membranes
* Cervical dilation > 4 cm
* Vaginal bleeding
* Major fetal abnormalities that are known at time of admission

Sex: Female
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A. Macones, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States